CLINICAL TRIAL: NCT05473065
Title: A Prosthetic Foot Test-Drive Strategy for Improving Stability and Falls-Related Outcomes in Veterans With Leg Amputations
Brief Title: A Prosthetic Foot Test-Drive Strategy for Improving Stability in Veterans With Leg Amputations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: VA Puget Sound Health Care System (U.S. Federal Agency); Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency); University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: W81XWH-20-1-0291; MD15 (Other Grant/Funding Number: Seattle Institute for Biomedical and Clinical Research); CDMRP-OP190048 (Other: DoD Congressionally Directed Medical Research Programs)
Record Dates: First submitted 2022-06-23; First posted 2022-07-25 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Amputation
Keywords: amputation; rehabilitation; balance; stability; falls; emulator; prosthetics

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be blinded to the commercial prosthetic foot type and to the emulated foot condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Multiaxial Prosthetic Foot Emulator (PFE) (Experimental): The multiaxial Prosthetic Foot Emulator (PFE) is a customizable robotic prosthetic foot that can mimic commercial feet to predict how prosthesis users will respond to candidate feet. Participants will walk with the PFE using three different modes (emulating three commercial feet) under different walking conditions.
  Interventions: Device: Multiaxial Prosthetic Foot Emulator
- Commercially available prosthetic feet (Active Comparator): Participants will walk under different walking conditions using three different commercial prosthetic feet.
  Interventions: Device: Commercially available prosthetic feet

INTERVENTIONS:
Device: Multiaxial Prosthetic Foot Emulator — Participants will walk in the laboratory with the multiaxial Prosthetic Foot Emulator (PFE) in three foot modes corresponding to commercial prosthetic study feet. Walking conditions will include self-selected comfortable, slow, and fast speeds, inclines, cross slopes, and uneven terrain.
  Arms: Multiaxial Prosthetic Foot Emulator (PFE)
Device: Commercially available prosthetic feet — Participants will walk in the laboratory with the commercial prosthetic study feet in three foot modes corresponding to commercial prosthetic study feet. Walking conditions will include self-selected comfortable, slow, and fast speeds, inclines, cross slopes, and uneven terrain.
  Additionally, participants will be fit with one of the commercial prosthetic study feet and wear it at home and in the community for approximately one week. Participants will return to the laboratory to follow-up testing, and will complete the community trial with each of the three commercial prosthetic study feet.
  Arms: Commercially available prosthetic feet

SUMMARY:
Objective/Hypotheses and Specific Aims: The first aim of this proposal is to determine the effects of commercial prosthetic feet of varying stiffness on stability and falls-related outcomes in Veterans with TTA. The second aim is to determine whether a PFE can be used to predict stability and balance-confidence outcomes with corresponding commercial prosthetic feet. The third and final aim is to determine whether a brief trial of commercial prosthetic feet can predict longer-term stability and balance-confidence outcomes in Veterans with TTA.

Study Design: The investigators will use a participant blinded cross-over study with repeated measurements in Veterans and Service members with TTA. Up to 50 participants will be enrolled at each of the two study sites VA Puget Sound and VA Minneapolis. Participants will complete up to 6 visits. After an initial assessment visit, participants will be assigned to the 'high' or 'low' mobility group, and then during visit 2 they will be randomized to use the PFE in three foot modes or the three corresponding actual (commercially available) feet during walking tests on difference surfaces in the laboratory (cross-slopes, inclines, even, and uneven ground). During visit 3 participants will repeat the procedures in the other condition (e.g., PFE if visit 2 included actual feet testing). At the end of visit 3 participants will be fit with one of the actual feet and wear it at home and in the community for approximately one week. At visit 4 participants will be fit with the next actual foot and repeat the 1 week use window. The same process will be followed for the final foot at visit 5, and the study foot will be returned at visit 6.

DETAILED DESCRIPTION:
Using a prosthesis allows many who experience lower leg amputation to regain functional abilities, but walking may be more difficult, and people with limb loss suffer from a wide range of mobility limitations including balance and stability impairments. Selecting an optimal prosthetic foot is an important aspect of maximizing mobility, limiting falls, and the achievement of functional goals for people with lower leg amputation (LLA), however there is limited evidence to guide this process. The current prosthetic prescription process relies on clinician experience and typically does not allow people with a leg amputation to easily try out different prosthetic feet. The investigators have developed a customizable robotic prosthetic foot that can mimic the mechanical properties of commercially available prosthetic feet in the coronal and sagittal planes without physically changing feet. This multiaxial 'prosthetic foot emulator' (PFE) can be attached to the prescribed prosthetic socket and worn like a regular prosthetic foot within the laboratory or clinic, providing people with LLA the opportunity to quickly 'test-drive' many prosthetic foot designs within a single test session. Trial and error with actual commercial prosthetic feet can be inefficient given the time and expense required for the purchasing and fitting of prosthetic feet. The PFE could provide a means to explore a range of feet over uneven, incline, and cross sloped surfaces in a very short period of time. This study aims to optimize stability and balance-related outcomes, to minimize falls, and to optimize vocational and avocational participation and functional quality for life for Veterans with LLA. This study will determine the effects of coronal and sagittal plane commercially-available prosthetic foot stiffness on stability and falls related outcomes and will evaluate the use of a test-drive strategy using a PFE to predict stability and balance-confidence outcomes with corresponding commercial prosthetic feet. Results from this study may contribute to increased understanding of how a patient-centered strategy for optimizing prosthetic prescription can improve patient satisfaction, functional outcomes, and balance confidence for Veterans and others with LLA.

ELIGIBILITY:
Inclusion Criteria:

* has a unilateral (one leg) transtibial (below-knee) amputation
* has used a prosthetic limb for walking for at least six months
* has a comfortably fitting prosthetic socket
* has a removable prosthetic foot attachment (i.e., is not rigidly attached to the back of the socket) so it can be used with study prosthetic feet
* be able to walk with a prosthetic limb sufficiently to participate in the experiment walking trials

Exclusion Criteria:

* contralateral limb or upper limb amputation that would interfere with completion of study activities
* are unable to use more than one of the test feet for any reason (e.g., excessively long residual limb that is not compatible with wearing study prosthetic feet)
* unable to walk under the minimal necessary study walking conditions in order to complete the study procedures without undo stress
* current surgical, neurological, rheumatologic, or lower limb musculoskeletal problem that significantly impairs ambulation (e.g., current ulcer, terminal illness)
* weight greater than 263lbs.
* inadequate cognitive or language function to consent to participate
* currently incarcerated
* impaired decision-making ability or the use of a legally authorized representative

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Self-report: perceived stability | Administered at baseline and during follow up testing with the commercial feet (approximately 2 hours)
  Correlation between prosthetic foot sagittal and coronal plane stiffness properties and perceived stability during walking on uneven ground and cross-slopes
Biomechanical measures: Medial/Lateral Margin of Stability (MOS) | Administered during follow up testing with the commercial feet (approximately 2 hours)
  Correlation between prosthetic foot sagittal and coronal plane stiffness properties and Medial/Lateral Margin of Stability (MOS) during walking on uneven ground and cross-slopes
Performance-based outcomes: Narrowing Beam Walking Test | Administered at baseline with the commercial feet (approximately 2 hours)
  Correlation between prosthetic foot sagittal and coronal plane stiffness properties and Narrowing Beam Walking Test score.
Performance-based outcomes: Narrowing Beam Walking Test | Administered during follow up testing with the commercial feet (approximately 2 hours)
  Correlation between prosthetic foot sagittal and coronal plane stiffness properties and Narrowing Beam Walking Test score.
Performance-based outcomes: Four Square Step Test | Administered at baseline with the commercial feet (approximately 2 hours)
  Correlation between prosthetic foot sagittal and coronal plane stiffness properties and Four Square Step Test score.
Performance-based outcomes: Four Square Step Test | Administered during follow up testing with the commercial feet (approximately 2 hours)
  Correlation between prosthetic foot sagittal and coronal plane stiffness properties and Four Square Step Test score.
Self-report: balance confidence Activities-specific Balance Confidence | Administered at baseline with the commercial feet (approximately 2 hours)
  Correlation between prosthetic foot sagittal and coronal plane stiffness properties and Activities-specific Balance Confidence (ABC) score
Self-report: Activity Restriction PROMIS Ability to Participate in Social Roles and Activities (APSRA) | Administered at baseline with the commercial feet (approximately 2 hours)
  Correlation between prosthetic foot sagittal and coronal plane stiffness properties and PROMIS Ability to Participate in Social Roles and Activities (APSRA)
Self-report: Activity Restriction PROMIS Ability to Participate in Social Roles and Activities (APSRA) | Administered during follow up testing with the commercial feet (approximately 2 hours)
  Correlation between prosthetic foot sagittal and coronal plane stiffness properties and PROMIS Ability to Participate in Social Roles and Activities (APSRA)
Self-report: perceived stability with emulated feet and commercial feet | Administered during initial testing with emulated and actual prosthetic feet (approximately two hours)
  Correlation between participants self-report perceived stability using the multiaxial prosthetic foot emulator and the commercial prosthetic study feet
Self-report: perceived stability with emulated feet and balance confidence using corresponding commercial feet | Administered during initial testing with emulated feet (approximately two hours)
  Correlation between participants self-report perceived stability using the multiaxial prosthetic foot emulator during initial testing and their balance confidence using the Activities-specific Balance Confidence during follow up with the corresponding commercial prosthetic foot
Self-report: perceived stability with emulated feet and balance confidence using corresponding commercial feet | Administered at follow up using the actual prosthetic feet (approximately two hours)
  Correlation between participants self-report perceived stability using the multiaxial prosthetic foot emulator during initial testing and their balance confidence using the Activities-specific Balance Confidence during follow up with the corresponding commercial prosthetic foot
Self-report: perceived stability with emulated feet and performance-based measures of stability (NBWT and FSST) using corresponding commercial feet | Administered during initial testing with emulated feet (approximately two hours)
  Correlation between participants self-report perceived stability using the multiaxial prosthetic foot emulator during initial testing and their performance-based stability using the Narrowing Beam Walking Test (NBWT) and Four Square Step Test (FSST) during follow up with the corresponding commercial prosthetic foot
Self-report: perceived stability with emulated feet and performance-based measures of stability (NBWT and FSST) using corresponding commercial feet | Administered at follow up using the actual prosthetic feet (approximately two hours)
  Correlation between participants self-report perceived stability using the multiaxial prosthetic foot emulator during initial testing and their performance-based stability using the Narrowing Beam Walking Test (NBWT) and Four Square Step Test (FSST) during follow up with the corresponding commercial prosthetic foot
Self-report: initial perceived stability and follow-up perceived stability | Administered during initial testing with the actual feet (approximately two hours)
  Correlation between initial perceived stability with each actual foot (relative to other feet) and perceived stability with the corresponding foot at follow-up
Self-report: initial perceived stability and follow-up perceived stability | Administered at follow up using the actual prosthetic feet (approximately two hours)
  Correlation between initial perceived stability with each actual foot (relative to other feet) and perceived stability with the corresponding foot at follow-up
Self-report: initial perceived stability and follow-up performance-based based measures of stability | Administered during initial testing with actual feet (approximately two hours)
  Correlation between initial perceived stability with each actual foot (relative to other feet) and performance-based stability using the Narrowing Beam Walking Test (NBWT) and Four Square Step Test (FSST) during follow up with the corresponding commercial prosthetic foot
Self-report: initial perceived stability and follow-up performance-based based measures of stability | Administered at follow up using the actual prosthetic feet (approximately two hours)
  Correlation between initial perceived stability with each actual foot (relative to other feet) and performance-based stability using the Narrowing Beam Walking Test (NBWT) and Four Square Step Test (FSST) during follow up with the corresponding commercial prosthetic foot

CONTACTS AND LOCATIONS:
Overall Officials: David C Morgenroth, MD, Principal Investigator — VA Puget Sound Health Care System
Locations (2):
- United States (2):
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - VA Puget Sound Health Care System, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ho TK, Halsne EG, Koehler-McNicholas SR, Hansen AH, Sawers A, Caputo JM, Curran CS, Lloyd A, Cave J, Morgenroth DC. Assessing the effects of prosthetic foot stiffness and foot preference on stability, balance confidence, and satisfaction in transtibial prosthesis users: Protocol for a randomized, participant-masked crossover trial using a 'test-drive' strategy. PLoS One. 2025 Oct 22;20(10):e0334497. doi: 10.1371/journal.pone.0334497. eCollection 2025. PMID 41124130